CLINICAL TRIAL: NCT01417117
Title: The Effect of Diffusion Weighted Imaging Abnormalities on Outcomes in Patients With Spontaneous Intracerebral Hemorrhage
Brief Title: Effect of Ischemic Strokes on Recovery From Intracerebral Hemorrhages
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Collaborators: American Heart Association (Other); Rush University (Other)
Responsible Party: Principal Investigator, Rajeev K Garg, Assistant Professor of Neurological Sciences and Neurosurgery, Rush University Medical Center
Other Study IDs: 11011402
Record Dates: First submitted 2011-08-12; First posted 2011-08-16 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Hemorrhage; Intracerebral, Nontraumatic; Ischemic Strokes; Diffusion Weighted Imaging Lesions
Keywords: Intracerebral Hemorrhage; Ischemic Stroke; Diffusion Weight Imaging Abnormalities; Neurologic Outcome
MeSH Terms: conditions — Hemorrhage; Ischemic Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spontaneous Intracerebral Hemorrhage: Patients with primary intracerebral hemorrhage within 24 hours of admission diagnosed by non-contrast head computed tomography (CT)

SUMMARY:
Intracerebral hemorrhage (ICH) occurs when small arteries in the brain rupture due to weakening by age, high blood pressure, and/or elevated cholesterol. In addition to artery rupture, recent data suggests that patients with ICH are also at risk for developing occlusion of arteries during the acute phase, called ischemic strokes. Data suggests these ischemic strokes can negatively impact patient outcomes. Diffusion weighted imaging (DWI) is a sequence on Magnetic Resonance Imaging (MRI) that is a sensitive marker for ischemic strokes in the brain. In this proposal, our primary aim is examine prospectively the effect DWI abnormalities have on functional outcomes in patients with ICH. Our hypothesis is that the DWI abnormalities found on MRI of the brain lead to worse functional outcomes in patients with ICH

DETAILED DESCRIPTION:
Diffusion weighted imaging (DWI) is a sensitive method to assess for secondary ischemia in patients with acute brain injury. By comparing the outcomes of patients with and without DWI abnormalities, we would able to assess the impact these lesions have on functional recovery in patients with ICH. Since no direct therapies exist for this disease, DWI abnormalities may be a novel target for intervention to improve outcomes. If traditionally assessed functional outcomes are not affected by DWI, the mechanism behind these lesions would still warrant further evaluation and potential treatment. Detection of subclinical infarcts has emerged as a potential surrogate marker for subsequent risk of stroke, vascular dementia, and cognitive impairment. Furthermore, the cause behind DWI lesions in acute ICH may lead to better understanding the pathophysiologic interplay between ischemic and hemorrhagic strokes.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years and < 80 years
* Spontaneous intracerebral hemorrhage documented by CT scan
* Less than 24 hours from time last seen normal to first medical evaluation
* No prior clinical history of stroke (i.e. subarachnoid hemorrhage, ICH, or ischemic strokes)

Exclusion Criteria:

* Pregnancy
* History of cancer
* Pre-admission mRS > 2
* Glasgow Coma Scale less than 5
* ICH secondary to aneurysm, vascular malformation, mycotic aneurysm, primary or metastatic tumor, trauma, warfarin-related ICH, acute-fibrinolytic associated ICH, or coagulopathy
* Associated epidural or subdural hematoma
* Surgical intervention < 48 hours from admission
* Hemodynamic instability (need for vasopressor therapy)
* Acute hypoxemic or hypercapnic respiratory failure
* History of deep venous thrombosis
* Contraindications to MRI based upon institutional safety checklist

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects for this study will be selected from patients admitted with a primary intracerebral hemorrhage to Rush University Medical Center's Neurosciences Intensive Care Unit.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2011-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | 3 months
  Modified Rankin Scale (mRS)

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale | 14 days or discharge
  National Institutes of Health Stroke Scale
Modified Rankin Scale (mRS) | 14 days
  Modified Rankin Scale (mRS)
Modified Rankin Scale (mRS) | 6 months
  Modified Rankin Scale (mRS)

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev K Garg, MD, Principal Investigator — Rush University Medical Center Deparment of Neurological Sciences
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No